CLINICAL TRIAL: NCT01407614
Title: Prevention of Secondary Ischemia After Aneurysmal Subarachnoid Hemorrhage With Cerebrospinal Fluid Drainage. A Randomized Controlled Trial
Brief Title: The Tilburg Vasospasm Study
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: patient enrollment too slow
Sponsor: Elisabeth-TweeSteden Ziekenhuis (Other)
Responsible Party: P.R.A.M. Depauw / drs, Neurosurgery St Elisabeth Hospital The Netherlands
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 15378
Record Dates: First submitted 2011-01-10; First posted 2011-08-02 (Estimated); Last update posted 2011-08-02 (Estimated); Status verified 2011-08

CONDITIONS: Brain Ischemia; Intracranial Vasospasm
Keywords: Subarachnoid hemorrhage; delayed cerebral ischemia; external lumbar drainage; vasospasm
MeSH Terms: conditions — Brain Ischemia; Vasospasm, Intracranial; Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- external lumbar drainage (Active Comparator): Within 96 hours of initial subarachnoid hemorrhage, patients were randomized for external lumbar drainage (ELD)of cerebrospinal fluid during a maximum of 7 days or standard treatment of subarachnoid hemorrhage without ELD
  Interventions: Procedure: external lumbar drainage (ELD) of cerebrospinal fluid
- No intervention (No Intervention): In this arm the patients received standard treatment following protocol for patients with subarachnoid hemorrhage

INTERVENTIONS:
Procedure: external lumbar drainage (ELD) of cerebrospinal fluid — Patients were randomized for external lumbar drainage of cerebrospinal fluid or standard treatment of a subarachnoid hemorrhage alone. External drainage was started within 96 hours of initial subarachnoid hemorrhage during 7 days at a maximum of 5-10 ml/hour.
  Arms: external lumbar drainage

SUMMARY:
In a prospective randomized controlled trial, the investigators aim to assess whether external lumbar drainage (ELD) of CSF is safe and reduces delayed cerebral ischemia and its sequelae in patients with an aneurysmal subarachnoid hemorrhage.

DETAILED DESCRIPTION:
Delayed cerebral ischemia (DCI) is a frequent complication after an aneurysmal subarachnoid hemorrhage (SAH). Its pathophysiological mechanism remains unclear but a role for cerebral vasospasm and the presence of blood in the arachnoid space is likely. A wash out of blood and blood breakdown products in the cerebrospinal fluid (CSF) could reduce the incidence of vasospasm and DCI.

We aim to assess whether external lumbar drainage (ELD) of CSF is safe and reduces secondary ischemia and its sequelae.

ELIGIBILITY:
Inclusion Criteria:

* spontaneous subarachnoid hemorrhage (SAH) with aneurysmal pattern graded as a Fisher grade III or higher on cerebral CT-scan.
* CSF drainage by external lumbar catheter can start within 96 hours after the initial SAH
* the drainage can start prior to the treatment of the ruptured aneurysm
* informed consent is signed by the patient or his representative

Exclusion Criteria:

* spontaneous SAH with aneurysmal pattern graded as a Fisher grade I or II on CT and perimesencephalic hemorrhages
* traumatic SAH
* symptomatic hydrocephalus on admission necessitating drainage (EVD or ELD)
* the presence of a large intraventricular bloodclot in the third or fourth ventricle on CT
* the presence of a mass lesion with significant cerebral midline shift
* all patients whose neurological condition is too poor to allow clinical recognition of signs and symptoms of cerebral vasospasm. This includes all patients with a Hunt and Hess Grade V who failed to improve after initial resuscitation
* no informed consent
* mycotic aneurysms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-12; Primary Completion 2009-03 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Clinical signs of delayed cerebral ischemia | Patients will be followed for the duration of admission, an expected average of 3 weeks
  DCI was diagnosed when all of the following criteria were met: (1) the onset of new neurological deficits such as confusion, disorientation, drowsiness, or focal deficit during post-hemorrhage days (4 to 14); (2) negative findings on CT obtained to rule out other causes of neurological deterioration such as hemorrhage, cerebral edema, or hydrocephalus. (3) No other identifiable cause of neurological deterioration such as hyponatriemia, hypoxia, drug toxicity, infection, or seizures.

SECONDARY OUTCOMES:
dichotomized Glasgow outcome score (GOS) | at discharge, an expected average of 3 weeks after initial bleeding
  Glasgow outcome scale was measured at discharge
new ischemic lesions on cerebral CT scan | at 3 months after initial bleeding
length of stay in intensive care unit | Patients will be followed from initial admission until discharge, an expected average of 3 weeks
  The length of stay in the intensive care unit will be measured.
rebleeding rate of unsecured aneurysms and complications of external lumbar drainage | Patients willl be followed from initial bleeding until treatment of aneurysm, an expected average of 3 days
  Evaluation of rebleeding rate of unsecured cerebral aneurysms during external lumbar drainage (ELD) of cerebrospinal fluid and evaluation of (other) complications of ELD such as (local)infection, discomfort/pain.
dichotomized Glasgow outcome score (GOS | at 3 months after initial bleeding
clinical signs of delayed cerebral ischemia | At 3 months after initial bleeding
  As stated in first primary outcome measure 'clinical signs of cerebral ischemia' during admission.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Depauw, MD, Principal Investigator — Elisabeth-TweeSteden Ziekenhuis
Locations (1):
- St Elisabeth Hospital, Tilburg, North Brabant, Netherlands